CLINICAL TRIAL: NCT06623903
Title: Early Breast Cancer, Endocrine Therapy Initiation, and Early Metabolic Health Changes: a Prospective Follow-up Study
Brief Title: Early Changes in Metabolic Health in Breast Cancer Patients Initiating Endocrine Therapy
Acronym: EMETA
Status: Not yet recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Signe Borgquist, Chair Professor, Senior Consultant, PhD, Aarhus University Hospital
Other Study IDs: 1-10-72-122-24; 09-2247 (Other Grant/Funding Number: The Danish Cancer Society)
Record Dates: First submitted 2024-09-27; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Early Breast Cancer; Metabolic Health; Estrogen Receptor Positive Breast Cancer
Keywords: Early breast cancer; Metabolic health; Endocrine therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — two blood samples analyzed for HbA1c, plasma glucose, hemoglobin, total cholesterol, triglycerides, LDL, HDL, and circulating estradiol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Early breast cancer patients initiating endocrine therapy: Patients with estrogen receptor-positive breast cancer initiating adjuvant endocrine therapy (either tamoxifen or aromatase inhibitors).

SUMMARY:
This clinical trial aims to investigate early metabolic health changes in early breast cancer patients that initiate antihormone therapy. Furthermore, how these changes are affected by estrogen level, treatment type, and patient characteristics. The hypothesis is, that initiation of antihormone therapy for early breast cancer patients is associated with an early deterioration in metabolic health after 3 months. This includes increased BMI (Body Mass Index), waist- and hip circumference, blood pressure, blood sugars, and lipids compared to when the patients initiate antihormone therapy. Concurrently, estradiol levels are expected to decrease. An estimated 112 patients initiating antihormone therapy at the Dept. of Oncology, Aarhus University Hospital (AUH) will be included in the study over 6 months from autumn 2024. Patients will have a metabolic screening on the day of initiating antihormone therapy and at 3-month antihormone treatment follow-up. The two metabolic screenings each consists of biometric measurements and a blood sample.

DETAILED DESCRIPTION:
Metabolic health, closely tied to overweight and type 2 diabetes, significantly influences disease risks, notably breast cancer. With over 2.5 billion overweight adults globally, the prevalence of associated health concerns is escalating. Breast cancer, the leading cause of female cancer-related mortality, is intricately linked to metabolic factors, including overweight and diabetes, particularly affecting estrogen receptor-positive tumors. Conversely, endocrine therapy as breast cancer treatment can exacerbate metabolic issues, increasing weight gain and the risk of type 2 diabetes. Despite its efficacy in reducing recurrence risk, endocrine therapy is associated with adverse metabolic effects, including elevated cholesterol levels. Estrogen, pivotal in metabolic homeostasis, remains poorly understood in the context of endocrine therapy and metabolic disruptions. This prospective study aims to elucidate this relationship, focusing on the initiation of endocrine therapy, metabolic health, and estradiol levels among early-stage breast cancer patients. Early breast cancer patients initiating endocrine therapy at Aarhus University Hospital from autumn 2024 and six months ahead will be extended an invitation for study participation, with immediate measurements. Metabolic health will be analyzed through weight, hip and waist circumference measurements, blood sugar, cholesterol, and estrogen at baseline and 3-month follow-up. Thorough data collection, including demographics, treatment modalities, and cancer characteristics, ensures a comprehensive understanding of this complex interplay. With 112 projected participants, this study aims to shed light on the intricate connections between endocrine therapy, patient characteristics, and metabolic health changes. Through this comprehensive approach, the investigators aim to enhance patient care and understanding of managing metabolic health alongside breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Invasive ER+ breast cancer
* No diabetes treatment
* Planned for initiation of any adjuvant endocrine therapy.

Exclusion Criteria:

* Pregnancy or lactation,
* Psychological, familial, sociological, or geographical conditions potentially hampering compliance with the study protocol and follow-up schedule; these conditions will be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early breast cancer patients consulted at Dept. of Oncology Aarhus University Hospital from autumn 2024 and 6 months ahead regarding adjuvant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic health changes | 3 months (from initiation of endocrine therapy to 3 month treatment follow-up)
  A change (deterioration or improvement) in metabolic health compared to baseline. Defined by a change in at least one of the below mentioned parameters.
Waist and hip circumference | 3 months (from initiation of endocrine therapy to 3 month treatment follow-up)
  A change in waist- and hip circumference compared to baseline
Blood pressure | 3 months (from initiation of endocrine therapy to 3 month treatment follow-up)
  A change in blood pressure compared to baseline
HbA1c | 3 months (from initiation of endocrine therapy to 3 month treatment follow-up)
  A change in circulating levels of glycated hemoglobin (HbA1c)
Cholestrerol | 3 months (from initiation of endocrine therapy to 3 month treatment follow-up)
  A change in blood cholesterol compared to baseline
Triglycerides | 3 months (from initiation of endocrine therapy to 3 month treatment follow-up)
  A change in triglycerides compared to baseline
LDL | 3 months (from initiation of endocrine therapy to 3 month treatment follow-up)
  A change in low-density lipoprotein (LDL) compared to baseline.
HDL | 3 months (from initiation of endocrine therapy to 3 month treatment follow-up)
  A change in and high-density lipoprotein (HDL) compared to baseline
Body Mass Index | 3 months (from initiation of endocrine therapy to 3 month treatment follow-up)
  A change in Body Mass Index (Height and weight combined, kg/m2)

SECONDARY OUTCOMES:
Estrogen level | 3 months (from initiation of endocrine therapy to 3 month treatment follow-up)
  Changes in circulating estrogen compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Signe Borgquist, Clinical Chair Professor, Ph.D, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Oncology, Aarhus University Hosptial, Aarhus N, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No